CLINICAL TRIAL: NCT03279354
Title: A Randomized Controlled Trial of the Effectiveness of a Smartphone Parent-child Partner Exercises Application on Enhancing Health-related Quality of Life of Children From Low-income Families
Brief Title: Smartphone Parent-child Partner Exercises Application Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW17-179
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Physical Activity
Keywords: Health-related quality of life; Physical activity; Smartphone application
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Family Move app intervention
  Interventions: Behavioral: Family Move app intervention
- Control group (Placebo Comparator): "HK FitNuts" app intervention
  Interventions: Behavioral: "HK FitNuts" app intervention

INTERVENTIONS:
Behavioral: Family Move app intervention — All the recruited parent-child pairs will be randomized after baseline assessment by an independent statistician using computer randomization tool to either the FAMILY MOVE app intervention group or the HK FitNuts app control group with a 1:1 allocation ratio. Although both groups receive a stand-alone app, the apps have distinct design features: use of competition and point elements (FAMILY MOVE app) or use of traditional demonstration elements (HK FitNuts app). After both groups have completed the 8-week intervention study and follow up measurements at 1 month, 6 months and 12 months after intervention, the control group will receive the same FAMILY MOVE app. Outcome assessments will be conducted by a trained interviewer blinded to the subject group allocation.
  Arms: Intervention group
Behavioral: "HK FitNuts" app intervention — The parent-child pairs in the control group will be given a link to download the "HK FitNuts" app which was developed by Hong Kong Association of Sports Medicine and Sports Science, Department of Orthopaedics & Traumatology of the Chinese University of Hong Kong and Hong Kong Dietitians Association to promote healthy lifestyle in Hong Kong. The app includes short video clips demonstrating basic individual exercise moves and provides other textual information related to PA. However, it does not have push notification function. In order to ensure that the intervention and control group will receive equal attention from our research team, we shall send a text about HK FitNuts and general exercise information to participants in the control group three times per week. Same as participants in the intervention group, the control group will also be asked to provide their weekly app usage and PA pattern by completing an online log at the end of each intervention week.
  Arms: Control group

SUMMARY:
Building upon our previous groundwork including the development of the FAMILY MOVE app and the pilot study, we will further evaluate the effectiveness of a simple parent-child partner exercise programme delivered by our FAMILY MOVE app on children's health-related quality of life through a single blinded randomized placebo-controlled trial (RCT). This RCT will sample 286 low-income parent-child pairs recruited from low income families in the community. Study participants will be randomized after baseline assessment by an independent statistician using computer randomization tool with 1:1 allocation ratio to either the FAMILY MOVE app intervention group or the HK FitNuts app control group. After both groups have completed the intervention study and follow up measurements at 1 month, 6 months and 12 months after intervention, the control group will receive the same FAMILY MOVE app. Outcome assessments will be conducted by a trained interviewer blinded to the subject group allocation at baseline, 1 month, 6 months and 12 months after intervention.

DETAILED DESCRIPTION:
The health benefits of regular physical activity (PA) are well recognized. An active lifestyle benefits health-related quality of life (HRQoL) through its effect on physical and mental health. Adults and children who regularly participate in PA reported better health-related quality of life (HRQoL) compared to those who do not. HRQoL is a multidimensional construct that captures the impact of illness on the person's ability to live a fulfilling life. Physical, social and psychological functioning are the most important domains of HRQoL in adults and children. Although many individuals realize the beneficial effects of PA, some lack motivation to sustain the recommended workout levels whilst others lack the means.

Physical activity to promote HRQOL In particular, parents living on a low income face a number of practical barriers such as unaffordable cost, lack of childcare support and limited time after work to engage in PA. Inactive parents will have difficulty to set PA examples and standards for their children. The amount of time they spend with children in activities together is also limited. Community programmes on parent-child partner exercises have the potential to enhance HRQoL in both parents and children by increasing their PA level and quality parent-child interactions. However, engaging low-income adults and children in PA programmes is challenging because of their busy schedule and limited access to PA facilities. Ubiquitous technologies such as web-based programme and smartphone applications (apps) may overcome the barriers to PA interventions for this difficult-to-reach population. Exercises for these families need to be simple and practical. The introduction of basic partner stretching and strength exercises that requires the parents and their children to help each other could be a good start for inactive families to change toward an active lifestyle. In addition to improved fitness, the shared joy and support during parent-child partner exercises may promote positive moods and better life satisfaction, i.e. HRQoL.

Mobile technology to promote PA Mobile device usage is rapidly increasing and half of the worldwide mobile phone subscriptions are in the Asia Pacific region. Advanced mobile devices such as smartphones are equipped with features of personal computer operating system such as persistent network connectivity and downloadable apps. Smartphone apps that combine textual information with gaming elements such as competition, scoreboard and point are growing in popularity as health promoting tools. These gaming elements harness people's aversion of losses which motivate them to keep doing exercises to achieve activity goals. In addition, apps also enable users to monitor, record and reflect on their behaviour and lifestyle in a more convenient and less stigmatizing way than traditional health interventions. However, their effectiveness in low-income families especially on HRQoL in children is unknown. Furthermore, most of the available apps are produced in Western populations and in English, which limit their applicability to low-income Chinese families. The few PA promotion apps that are available in Chinese language mainly target at individual adult users without considering whether the exercise moves are appropriate for children, which make it difficult to use in family intervention.

Previous work done by the research team Since 2012, our research team, in collaboration with a philanthropic foundation in Hong Kong (Kerry Group Foundation (Hong Kong) Limited (KGKF)), has provided various health empowerment interventions and comprehensive health assessment to a group of low income families in Hong Kong (166 low-income families from Tung Chung and 205 families with similar socio-demographic background from other districts of Hong Kong). We found that local Chinese adults from low-income families had poorer HRQoL than the general population [14]. Their children also had poorer HRQOL and more behavioral problems [15]. Results of our preliminary analysis showed that both parents and children from low-income families reported lower levels of PA per week than the recommended levels by World Health Organization (WHO). There was a positive correlation (r=0.25, p=0.001) between the total weekly time of physical activities (including walking, moderate-intensity or/and vigorous-intensity activities) in parents and children. Moreover, we delivered a pilot parent-child exercise course in October-November 2016 and found a significant gain of 12.5 points in the scores of Mental Health scale of Child Health Questionnaire - Parent Form - 50 (CHQ-PF50) of participating children. Our research team is working towards delivering this parent-child partner exercise programme as a smartphone app.

The development of the smartphone app on simple parent-child partner exercises, which is funded by a philanthropic foundation in Hong Kong (Kerry Group Foundation (Hong Kong) Limited (KGKF)) is currently in progress.

After expert consultation and review of relevant literature, we are developing a smartphone app "FAMILY MOVE" in Chinese language with the following features:

* Account login with a unique, anonymous participant number for each user family which would allow us to keep record of the user's frequency and duration of use of our app
* A fully automated 8-week parent-child partner exercise programme (release of Level 1 moves in Week 1-2; Level 2 moves in Week 3-4; Level 3 moves in Week 5-6; revision of all moves in Week 7-8) for young children aged 6 to 10 years and adolescents aged 11 years or above, respectively
* Each level consists of one warm-up clip (1 minute), 4 short exercise move demonstration clips with audio instructions (30 seconds per clip), and 1 long dance clip (3 minutes) integrating the four exercise moves with background music
* Points will be given to users after they have viewed an exercise move video clip. More points would be awarded to more difficult moves
* The scoreboard will display personal score as well as the scores of the top 5 users
* Three push notifications per week as prompts to motivate users to keep doing exercises

The exercise moves that the parent and children practiced in the pilot exercise course had been filmed after modification based on opinions from PA experts and would be used as demonstration videos in the app.

A pre-post pilot study will be conducted in 2017 on 166 parent-child pairs recruited from the group of families living in Tung Chung district in our cohort after the FAMILY MOVE app is produced. Parents of eligible families will be notified by SMS ("Short Message Service") and asked whether they agree or not to receive the FAMILY MOVE app as part of our health empowerment study. Parents who agree to participate in this pilot 8-week intervention study will be asked to complete the same set of questionnaires on their own HRQOL, PA levels and mental health condition and their children's HRQOL, behavior and PA levels at each assessment time point (baseline, 1-month and 6-month post intervention).

Building upon such groundwork and existing evidence, in the present study our team would like to evaluate further by launching a randomized-controlled trial (RCT) examining the effectiveness of a simple parent-child partner exercise programme delivered as a smartphone app "FAMILY MOVE" in enhancing the HRQoL and PA level of children from low-income families.

Aims and Hypotheses to be Tested:

Study Objectives

1. To evaluate the effectiveness of the smartphone app "FAMILY MOVE" in improving the HRQoL of children;
2. To evaluate the effectiveness of the smartphone app "FAMILY MOVE" in improving the PA levels of children;
3. To explore the associations between "FAMILY MOVE" app usage and HRQoL and PA of children.

Study hypotheses

1. Compared to the control group, children from the intervention group will show better HRQoL (measured by the Psychosocial Summary scores of the Child Health Questionnaire - Parent Form - 50 (CHQ-PF50)) at 1 month, 6 months and 12 months after intervention.
2. Compared to the control group, children from the intervention group will show greater PA measured by the METS (Metabolic Equivalent for Task) -minutes/week at 1 month, 6 months and 12 months after intervention.
3. There is a positive correlation of improvement in HRQoL and PA levels of children with the time they spend on the FAMILY MOVE app.

ELIGIBILITY:
Inclusion Criteria:

* Family monthly household income does not exceed 75% of Hong Kong's median monthly household income at enrollment;
* Family has at least one parent and one child aged 7 to16 years at enrollment;
* At least one parent has a smartphone with iOS or Android mobile operating system.

Exclusion Criteria:

* Both parents and children cannot understand or read traditional Chinese
* Parents or children with a medical condition limiting ability to exercise
* Previous use of the apps of interest

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Child Psychosocial Health at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  Chinese Child Health Questionnaire - Parent Form - 50 (CHQ-PF50); including 12 domain scales (General Health, Physical Functioning, Role/Social Limitations - Emotional/Behavioral, Role/Social Limitations - Physical, Bodily Pain/Discomfort, Behavior, Mental Health, Self-Esteem, Parental Impact - Emotion, Parental Impact - Time, Family Activities, and Family Cohesion) and 2 summary scores (Physical Summary Score and Psychosocial Summary Score). Higher scores indicate better HRQoL.
Change from Baseline Child Total Physical Activity Score (MET-minutes/week) at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  International Physical Activity Questionnaire - Short Form - Chinese version (IPAQ-SF); including seven questions on the frequency and duration of time spent in physical activity in the past 7 days to calculate a score for each domain (walking, moderate-intensity activities and vigorous-intensity activities) and an overall grand total expressed in MET-minutes/week.

SECONDARY OUTCOMES:
Change from Baseline Parental Mental and Physical Health at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  Chinese (Hong Kong) translation of 12-item Short-Form Health Survey-version 2 (SF-12v2); a generic HRQoL measure including 8 domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) and two (mental health and physical health) summary scores.
Change from Baseline Child SDQ Total Difficulties Scores at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  Chinese Strength and Difficulties Questionnaire (SDQ); including 5 subscales of emotional symptoms, conduct problems, hyperactivity/inattention, prosocial behaviors and peer relationship problems. Higher scores indicate worse behavior for all except the prosocial behavior score. The scores of the four subscales that measure symptoms or problems can be summated to a total difficulties score
Change from Baseline Parent Total Physical Activity Score (MET-minutes/week) at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  International Physical Activity Questionnaire - Short Form - Chinese version (IPAQ-SF); including seven questions on the frequency and duration of time spent in physical activity in the past 7 days to calculate a score for each domain (walking, moderate-intensity activities and vigorous-intensity activities) and an overall grand total expressed in MET-minutes/week.
Change from Baseline Parental DASS scores on each subscale (Depression, Anxiety and Stress) at 1 month and 6 month post intervention | baseline, 1 month, and 6 month post intervention
  Chinese Depression Anxiety Stress Scale - 21 (DASS - 21); including 3 subscales, each with 7 items rating the severity/frequency of anxiety symptoms, depression symptoms, and stress respectively

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Lo Kuen Lam, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wong RSM, Yu EYT, Wong TW, Fung CSC, Choi CSY, Or CKL, Liu KSN, Wong CKH, Ip P, Lam CLK. Development and pilot evaluation of a mobile app on parent-child exercises to improve physical activity and psychosocial outcomes of Hong Kong Chinese children. BMC Public Health. 2020 Oct 14;20(1):1544. doi: 10.1186/s12889-020-09655-9. PMID 33054753
- See also: Development of a mobile on parent-child exercies — https://doi.org/10.1186/s12889-020-09655-9